CLINICAL TRIAL: NCT00636701
Title: Improving Rehabilitation by Magnetic Brain Stimulation: Improving Motor Recovery After Stroke
Brief Title: Improving Rehabilitation by Magnetic Brain Stimulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B4657-P
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primed rTMS (Experimental): Receive 10 min. of 6-Hz rTMS Repetitive Transcranial Magnetic Stimulation at 90% RMT (3,600 pulses). Followed by 30 min. of 1-Hz rTMS at 95% RMT (1,880 pulses)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Unprimed rTMS) (Placebo Comparator): Receive 10 min. of sham rTMS Repetitive Transcranial Magnetic Stimulation. Followed by 30 min. of 1-Hz rTMS at 95% RMT (1,880 pulses)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — We will position a coil over the motor cortex of the head and give a series of stimulations (called magnetic pulses).
  Other Names: RTMS

SUMMARY:
We hope to understand the properties of the motor cortex in the brain of people with stroke using non-invasive magnetic stimulation.

DETAILED DESCRIPTION:
This case series assesses the effects of five consecutive days of low-frequency (1 Hz) repetitive transcranial magnetic stimulation (rTMS) with and without a 6-Hz primer. Although this paper studies able-bodied individuals, similar rTMS protocols are used to facilitate motor recovery in patients with hemiplegia following stroke. However, the cortical mechanisms associated with repeated daily doses of rTMS are not completely understood.

ELIGIBILITY:
Inclusion Criteria:

* 3-24 months post stroke
* upper limb paresis
* CES-D below 16,

Exclusion Criteria:

* history of seizure
* metal in head
* score of less than 24 on the Folstein Mini-Mental Status Exam
* clinical judgement of excessive frailty or lack of stamina (e.g. cannot attend to instructions, stay awake, engage in functional activities)
* serious uncontrolled medical condition
* excessive pain in any joint of the more affected extremity that could limit ability to cooperate with the intervention as judged by the examining clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Butler, PhD MS BA, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- [Result] Glielmi CB, Butler AJ, Niyazov DM, Darling WG, Epstein CM, Alberts JL, Hu XP. Assessing low-frequency repetitive transcranial magnetic stimulation with functional magnetic resonance imaging: a case series. Physiother Res Int. 2014 Jun;19(2):117-25. doi: 10.1002/pri.518. Epub 2011 Jul 18. PMID 21766399

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Receive rTMS (Repetitive Transcranial Magnetic Stimulation)
  Repetitive Transcranial Magnetic Stimulation: We will position a coil over the motor cortex of your head and give a series of stimulations (called magnetic pulses) for 2 minutes
- Arm 2: Receive sham rTMS (Repetitive Transcranial Magnetic Stimulation)
  Repetitive Transcranial Magnetic Stimulation: We will position a coil over the motor cortex of your head and give a series of stimulations (called magnetic pulses) for 2 minutes
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage BOLD (Blood-oxygen-level Dependent Contrast Imaging) Signal From Baseline at 2 Weeks
Description: Blood-oxygen-level dependent contrast imaging, or BOLD-contrast imaging, is a method used in functional magnetic resonance imaging (fMRI) to observe different areas of the brain or other organs, which are found to be active at any given time. In 1990, three papers published by Seiji Ogawa and colleagues showed that haemoglobin has different magnetic properties in its oxygenated and deoxygenated forms, both of which could be detected using MRI. This leads to magnetic signal variation which can be detected using an MRI scanner. Given many repetitions of a thought, action or experience, statistical methods can be used to determine the areas of the brain which reliably have more of this difference as a result, and therefore which areas of the brain are active during that thought, action or experience. The percentage BOLD was measures at day 0 and day two weeks. We measured the change in the dependent measure from day 0 to day 2 weeks .
Time Frame: Baseline (day 0) and 2 weeks
Population: Four right-handed healthy volunteers (two men, aged 20-50 years) participated in a double-blind study of primed and unprimed rTMS.
Measure: Mean (Standard Deviation); unit: percentage change of BOLD
Groups:
- Number of Participants Who Received Primed rTMS: Number of participants who received 10 min. of 6-Hz rTMS Repetitive Transcranial Magnetic Stimulation at 90% RMT (3,600 pulses). Followed by 30 min. of 1-Hz rTMS at 95% RMT (1,880 pulses)
- Number of Participants Who Received Unprimed rTMS: Number of participants who received 10 min. of sham rTMS Repetitive Transcranial Magnetic Stimulation. Followed by 30 min. of 1-Hz rTMS at 95% RMT (1,880 pulses)
Arm/Group | Number of Participants Who Received Primed rTMS | Number of Participants Who Received Unprimed rTMS
Number analyzed (Participants) | 2 | 2
percentage change of BOLD | 3 (.5) | 2 (.25)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes